CLINICAL TRIAL: NCT06668532
Title: Longitudinal Well-Being Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Flourish Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Flourish2024-01
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: well-being; digital; positive psychology; students

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flourish app condition (Experimental): Participants in this condition will gain access to the Flourish app and be instructed to use it at least twice a week for 6 weeks.
  Interventions: Device: Digital toolkit
- Control Condition (Active Comparator): Participants in the control condition will gain access to mental health resources each week for 6 weeks and be instructed to reflect on how the information in the resources can be applied to their own lives.
  Interventions: Other: National mental health resources

INTERVENTIONS:
Device: Digital toolkit — Access to the Flourish app and instruction to use at least twice a week for 6 weeks.
  Other Names: Flourish app
  Arms: Flourish app condition
Other: National mental health resources — Access to national mental health resources from Mental Health America, which can be found here: https://mhanational.org/ten-tools. Participants will receive one resource each week for 6 weeks and each time, will be asked to reflect on how the information can be applied to their own lives.
  Other Names: Website links
  Arms: Control Condition

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the Flourish app-a digital toolkit providing science-based well-being practices-in enhancing mental health among students. The main questions it aims to answer are:

* Does regular use of the Flourish app improve well-being, emotional resilience, and stress management?
* Is more frequent use of the Flourish app associated with greater improvements in these outcomes?

Researchers will compare outcomes between participants using the Flourish app and a control group receiving curated national mental health resources to assess the app's impact.

Participants will:

* Complete an initial 15-minute survey to establish baseline mental health
* Those in the Flourish app condition will use the app at least twice weekly, while those in the control condition will receive weekly mental health resources and reflect on their application
* Complete biweekly follow-up surveys over six weeks, with a final survey three months later

ELIGIBILITY:
Inclusion Criteria:

* Currently a student
* Fluent in English
* No uncontrolled mental health condition that significantly impacts daily life
* Prolific approval rate within the 95-100% range
* Minimum of 20 previous Prolific submissions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Flourishing Scale | Baseline, 6 weeks post-baseline, and 3-month follow-up
  The Flourishing Scale (Diener et al., 2009) is an 8-item measure of psychological well-being. Respondents rate items from 1 ("Strongly disagree") to 7 ("Strongly agree"), yielding a total score range from 8 to 56. Higher scores indicate greater well-being and flourishing.
Depression (PHQ-8) | Baseline, bi-weekly for 6 weeks (3 time points), and 3-month follow-up
  The PHQ-8 is an 8-item measure assessing depression severity over the past two weeks. Each item scores from 0 ("not at all") to 3 ("nearly every day"), with total scores from 0 to 24. Higher scores indicate greater depression severity.
Anxiety (GAD-7) | Baseline, bi-weekly for 6 weeks (3 time points), and 3-month follow-up
  The GAD-7 (Generalized Anxiety Disorder-7) is a 7-item measure assessing anxiety severity. Each item is rated from 0 ("not at all") to 3 ("nearly every day"), with total scores ranging from 0 to 21. Higher scores indicate greater anxiety severity.
Perceived Stress (PSS-4) | Baseline, bi-weekly for 6 weeks (3 time points), and 3-month follow-up
  The PSS-4 (Perceived Stress Scale-4) is a 4-item measure of perceived stress, rated from 0 ("never") to 4 ("very often"). Scores range from 0 to 16, with higher scores indicating greater stress.
Subcomponents of Affect Scale | Baseline, bi-weekly for 6 weeks (3 time points), and 3-month follow-up
  The Subcomponents of Affect Scale (SAS) is an 18-item measure of affect, divided into nine positive and nine negative adjectives. Positive subscales include calm, well-being, and vigor, while negative subscales include depression, anxiety, and anger. Participants rate each adjective from 0 (not at all accurate) to 4 (extremely accurate) based on their feelings over the past two weeks. Total scores for positive and negative affect are summed from their subscales.
Resilience | Baseline, 6 weeks post-baseline, and 3-month follow-up
  The Brief Resilience Scale (BRS; Smith et al., 2008) is a 6-item measure of stress recovery, rated from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate a stronger ability to "bounce back" after setbacks.

SECONDARY OUTCOMES:
Loneliness | Baseline, 6 weeks post-baseline, and 3-month follow-up
  The UCLA 3-Item Loneliness Scale is a brief measure assessing subjective feelings of loneliness and social isolation. Participants rate each item on a 3-point scale, from 1 (hardly ever) to 3 (often), with higher scores indicating greater loneliness.
Social Fit | Baseline, 6 weeks post-baseline, and 3-month follow-up
  The Sense of Social Fit Scale (Walton & Cohen, 2007) measures students' perceived belonging within their school environment. For our purposes, we used a shortened version with two items: "I fit in well at my school" and "Other people understand more than I do about what is going on at my school," rated on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree).
Perceived Cohesion | Baseline, 6 weeks post-baseline, and 3-month follow-up
  The Perceived Cohesion Scale (Bollen & Hoyle, 1990) measures a sense of belonging and morale within a community using a Likert scale from 0 (strongly disagree) to 10 (strongly agree). For our purposes, we use a single-item version: "I see myself as part of the campus community."
Expectations and Experiences of Chatbots | Baseline, 6 weeks post-baseline, and 3-month follow-up
  This measure, adapted from the Working Alliance Inventory - Short Revised (WAI-SR), assesses participants' expectations and experiences with chatbots. Participants rate anticipated and actual interactions across three areas-Goal, Task, and Bond-on a 5-point scale from 1 (seldom) to 5 (always), with higher scores indicating stronger alignment.
Multi-Dimensional Measure of Trust | 6 weeks post-baseline, and 3-month follow-up
  The Multi-Dimensional Measure of Trust (MDMT; Ullman & Malle, 2023) assesses perceived trustworthiness of the Flourish chatbot, Sunnie, through a set of 10 attributes (Form A), rated from 0 (Not at all) to 5 (Very), with a 'Does Not Fit' option. Only participants in the Flourish app condition complete this measure.
Academic Self Efficacy | Baseline, 6 weeks post-baseline, and 3-month follow-up
  The Academic Self-Efficacy scale (van Zyl et al., 2022) measures students' confidence in their ability to succeed academically. Participants rate their agreement with statements such as "I generally manage to solve difficult academic problems if I try hard enough" on a 5-point scale, from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate greater self-belief in tackling academic challenges and achieving study-related goals.
School Perceptions | Baseline, 6 weeks post-baseline, and 3-month follow-up
  School perceptions are measured using two single-item measures from the Healthy Minds Survey, along with an adapted Inclusion of Other in the Self (IOS) scale to capture closeness to the university.
  The first item rates agreement with the statement, "At my school, students' mental and emotional well-being is a priority," on a scale from 1 (strongly agree) to 6 (strongly disagree).
  The second item rates satisfaction with the overall school experience from 1 (very dissatisfied) to 6 (very satisfied).
  For university closeness, participants select one image from a series of overlapping circles that best represents their relationship with the university, with greater overlap indicating a stronger connection.

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified participant data on OSF from each study timepoint across both conditions, including all data used in our analyses.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning upon submission for publication with no end date.